CLINICAL TRIAL: NCT06541002
Title: Multi-Site Randomized Controlled Trial of a Novel Digital Application (SHIFT) to Improve Outcomes for Hematopoietic Stem Cell Transplant Survivors
Brief Title: A Novel Digital Application (SHIFT) to Improve Outcomes for Hematopoietic Stem Cell Transplant Survivors
Acronym: SHIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-256; 1R01CA282182-01 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sexual Dysfunction; Stem Cell Transplant Complications; Bone Marrow Transplant Complications
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHIFT Intervention Group (Experimental): SHIFT is a self-administered, multi-component digital application for HCT survivors, incorporating several features to promote engagement and health behavior change, and includes gamification strategies, videos of HCT survivors, intimacy exercises, and optional content.
  Interventions: Behavioral: SHIFT Intervention Group
- Enhanced Usual Care Group (Active Comparator): Patients assigned to enhanced usual care group will not receive access to the SHIFT application. They will meet with their HCT clinician and maybe referred to specialist care at the patients' request or at the discretion of the HCT clinician.
  Interventions: Behavioral: Enhanced Usual Care Group

INTERVENTIONS:
Behavioral: SHIFT Intervention Group — Participants assigned to SHIFT will meet with their HCT clinician for a brief medical examination to assess the need for medications for erectile dysfunction, vaginal atrophy, or genital graft-versus-host disease; and start using SHIFT at their desired pace over 8 weeks to complete five modules.
  Arms: SHIFT Intervention Group
Behavioral: Enhanced Usual Care Group — Participants assigned to the enhanced usual care group will meet with their HCT clinician for a brief medical examination to assess the need for medications for erectile dysfunction, vaginal atrophy, or genital graft-versus-host disease; and maybe referred to a psychologist, urologist, or gynecologist at the participants' request or at the discretion of the HCT clinician.
  Arms: Enhanced Usual Care Group

SUMMARY:
This research study is evaluating the efficacy of a novel self-administered digital application for improving sexual health outcomes, quality of life, and psychological distress in hematopoietic stem cell transplant survivors.

DETAILED DESCRIPTION:
Autologous and Allogeneic hematopoietic stem cell transplant (HCT) are potentially curative treatments for many patients with hematologic malignancies and benign hematologic conditions. The use of HCT has increased over the last decade. HCT survivors experience a substantial and drastic deterioration in their sexual function that persists for many years post-HCT. Sexual dysfunction is the most common long-term complication in HCT survivors. Sexual health problems have negative consequences on patients' quality of life (QOL) and mood, including the individual's identity and self-esteem, fatigue, relationship discord, intimacy problems, and distress. The etiology of sexual dysfunction in HCT survivors is multi-factorial, and can stem from biological, interpersonal, psychological, and social factors. Given the multi-factorial nature underlying sexual dysfunction in this population, a multimodal approach is required to address them. Clinicians lack sufficient training to address sexual health problems in HCT survivors. HCT survivors report having little communication with their clinicians about sexual health. HCT survivors would benefit from interventions to empower them to communicate with their clinicians about their sexual health.

Despite the well-documented burden of sexual dysfunction in HCT survivors, interventions tailored to address their unique sexual health concerns are lacking. Given the multi-factorial nature of sexual health concerns in HCT survivors, interventions must address these diverse needs, and should therefore ideally be addressed by a multidisciplinary team of sexual health experts, psychologists, gynecologists, and urologists. Although a few transplant centers have a multidisciplinary sexual health clinic, the lack of professionals trained in addressing sexual health concerns severely limits the dissemination of such a complex service model. In addition, HCT survivors often find it difficult to attend multiple clinic appointments and coordinate their care among various specialists. Limited availability of sexual health clinicians also hinders the scalability and dissemination of sexual health interventions to address the needs of HCT survivors. Digital health interventions can enhance access and broad dissemination of psychological and supportive care interventions and will enable patients to access the intervention in the privacy of their home given the sensitivity of the topic, engage their partners with the content, and avoid additional clinic visits. A successful evidence-based sexual health intervention was adapted to a digital app for HCT survivors. The active components of an in-person sexual health intervention for HCT survivors were leveraged to develop the self-administered digital application, Sexual Health and Intimacy Following Transplant (SHIFT) to address the sexual health concerns of HCT survivors. This multi-site randomized trial will test the efficacy SHIFT for improving sexual health outcomes, quality of life, and psychological distress in HCT survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years) who underwent autologous or allogeneic HCT > three months prior to study enrollment
* Screen positive for sexual health concerns causing distress based on the National Comprehensive Network (NCCN) survivorship guidelines screening questions

Exclusion Criteria:

* Patients who do not comprehend English or Spanish since SHIFT will only be available in these two languages for this efficacy trial.
* Patients with any major uncontrolled psychiatric disorder or other comorbid cognitive conditions, which the treating HCT clinician believes would prohibit the patients' capacity to provide informed consent and participate in study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Global satisfaction with sex at week 8 as measured by the global satisfaction with sex domain from the Patient-Reported Outcomes Measurement Information System (PROMIS) Satisfaction with Sex Life scale. | Week 8
  To compare patient global satisfaction with sex scores at week 8 after enrollment between those receiving SHIFT versus enhanced usual care as measured by the PROMIS global satisfaction with sex domain from the PROMIS Scale v2.0 Satisfaction with Sex Life.
  Higher scores indicate higher satisfaction with sex life, and lower scores indicate less satisfaction with sex life.

SECONDARY OUTCOMES:
Global satisfaction with sex (longitudinally) as measured by the global satisfaction with sex domain from the PROMIS Satisfaction with Sex Life scale | Up to week-24
  To compare patient global satisfaction with sex longitudinally between those receiving SHIFT versus enhanced usual care as measured by the global satisfaction with sex domain from the PROMIS Scale v2.0 Satisfaction with Sex Life scale.
  Higher scores indicate higher satisfaction with sex life, and lower scores indicate less satisfaction with sex life.
Sexual interest as measured by the interest in sexual activity domain from the PROMIS Sexual Function and Satisfaction scale | Up to week-24
  To compare sexual interest both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the interest in sexual activity domain from the PROMIS Scale v2.0 Sexual Function and Satisfaction scale.
  Higher scores indicate more interest, and lower scores indicate less interest.
Sexual function (orgasm) as measured by the by the Orgasm - Pleasure domain from the PROMIS Sexual Function and Satisfaction scale | Up to week-24
  To compare sexual function (orgasm) both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the Orgasm - Pleasure domain from the PROMIS Scale v2.0 - Sexual Function and Satisfaction scale.
  Higher scores from the Orgasm - Pleasure domain from the PROMIS Scale - Sexual Function and Satisfaction indicate more pleasurable orgasms.
Sexual function (vaginal discomfort, and vaginal lubrication) as measured by the Female Sexual Function Index scale | Up to week-24
  To compare sexual function (vaginal discomfort, and vaginal lubrication) both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the Female Sexual Function Index (FSFI) for female participants.
  Higher scores of FSFI indicate greater levels of sexual functioning and lower scores indicate lower levels of sexual functioning.
Erectile function as measured by the International Index of Erectile Function scale | Up to week-24
  To compare erectile function both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the International Index of Erectile Function (IIEF-5) for male participants.
  Higher scores of IIEF-5 indicate greater levels of sexual functioning and lower scores indicate lower levels of sexual functioning.
Quality of Life as measured by the Functional Assessment of Cancer Therapy- Bone Marrow Transplant scale | Up to week-24
  To compare quality of life (QOL) both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the Functional Assessment of Cancer Therapy- Bone Marrow Transplant (FACT-BMT) scale.
  Higher scores on FACT-BMT indicate better QOL.
Anxiety symptoms as measured by the Hospital Anxiety and Depression Scale | Up to week-24
  To compare anxiety symptoms both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the Hospital Anxiety and Depression Scale (HADS) Anxiety subscale.
  Lower scores on HADS anxiety subscale indicate less anxiety (score: 0-7-Normal, 8-10-Mild, 11-15-Moderate, 16-21-Severe).
Depression symptoms as measured by the Hospital Anxiety and Depression Scale | Up to week-24
  To compare depression symptoms both at week 8 and longitudinally after enrollment between those receiving SHIFT versus enhanced usual care as measured by the Hospital Anxiety and Depression Scale (HADS) Depression subscale.
  Lower scores on HADS depression subscale indicate absence of depression (score: 0-7-Normal, 8-10-Mild, 11-15-Moderate, 16-21-Severe).

OTHER OUTCOMES:
The proportion of participants who are sexually active using the PROMIS Sexual Activity Screener | Up to week-24
  To compare the proportion of participants who are sexually active between those receiving SHIFT versus enhanced usual care as measured by the PROMIS Sexual Function and Satisfaction (SexFS) Version 2.0: Screener.
Emotional and sexual intimacy as measured by the emotional and sexual intimacy subscales in Personal Assessment of Intimacy in Relationship scale | Up to week-24
  To compare emotional and sexual intimacy between those receiving SHIFT versus enhanced usual care using the emotional and sexual intimacy subscales from the Personal Assessment of Intimacy in Relationship (PAIR) emotional and sexual intimacy subscales.
  Lower scores indicate greater relationship intimacy, and higher scores indicate lower relationship intimacy.
To compare participants' self-efficacy for discussing sexual health with their transplant clinicians using the Self-Efficacy Questionnaire | Up to week-24
  To compare participants' self-efficacy for discussing their sexual health with their transplant clinician's between those receiving SHIFT versus enhanced usual care using the Self-Efficacy Questionnaire.
  This will be assessed using two items with score ranging from 0-20. Higher scores indicate better self-efficacy, and lower scores indicate lesser self-efficacy.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Miami, Coral Gables, Florida
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Mass General Brigham Innovation team
URL: https://www.massgeneralbrigham.org/en/research-and-innovation/innovation